CLINICAL TRIAL: NCT06619041
Title: Harnessing the Power of Social Support for Weight Management: a Randomized Controlled Trial of HealthyTogether
Brief Title: HealthyTogether: RCT of a Dyadic Weight Management Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 23-040
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Overweight
Keywords: Weight Loss; Weight Loss Programs; Social Support; Diet; Physical Activity; Virtual Medicine; Family; Dyadic
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Brief, virtual, dyadic weight management intervention
Who Masked: Outcomes Assessor
Masking Description: Study staff who measure the primary outcome (weight) and conduct other outcome assessments at 6-months will remain masked to the treatment arm assignment of participants throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Receives the brief, virtual, dyadic HealthyTogether weight management intervention in addition to usual care.
  Interventions: Behavioral: HealthyTogether
- Usual Care Arm (No Intervention): Receives a brief letter with information about weight management and couples/family resources in addition to usual care.

INTERVENTIONS:
Behavioral: HealthyTogether — HealthyTogether is a brief (8-session), virtual, dyadic weight management intervention.
  Arms: Treatment Arm

SUMMARY:
Four in five Veterans have overweight or obesity. However, few eligible Veterans achieve meaningful weight loss in VA's national MOVE! Weight Management Program. Family and friends strongly influence a person's health behaviors and weight. Including a close family member or friend in weight management may improve weight management outcomes. This study will test whether an 14-week, 8-session virtual weight management program that includes Veterans and a support person (e.g., family member or friend) leads to weight loss. The investigators will also test whether the program leads to improvements in weight-related health behaviors, including physical activity and diet, and relationship quality.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity is more than 80% among VA users, increasing risk of morbidity and mortality. In 2006, VA nationally implemented the MOVE! Weight Management Program, an evidence-based behavioral weight management program. Effectiveness of MOVE! is suboptimal: <20% of all participants and only 30% of those with intense and sustained participation achieve clinically meaningful weight loss. Furthermore, only 8-9% of eligible Veterans attend any MOVE! sessions and, among those who do, half attend only a single session. Taken together, <2% of the 3.2 million eligible Veterans lose clinically meaningful weight in MOVE!. Therefore, additional weight management approaches are needed to address obesity at the VA population-level.

One strategy to improve behavioral weight management effectiveness is by leveraging social relationships. Social support improves weight management program initiation, retention, and short and long-term weight loss and is also a major driver of weight-related behaviors, such as physical activity and diet quality. However, social relationships can also impede weight management, for example, when close others (e.g., family and friends) undermine or do not support behavior change. The key to addressing this double-edged sword of social relationships may be through dyadic approaches that include close others in behavioral weight management with a focus on improving communication and relationship quality.

HealthyTogether is a brief, virtual weight management program for Veterans and a close other ("partner"). Over 14 weeks, individual dyads receive 8 hour-long video sessions with a clinician. Session content includes physical activity, diet, and weight management medication education; goal setting; and relationship and communication skills training and practice, informed by evidence-based dyadic treatments. This study is a two-site hybrid type I effectiveness-implementation randomized controlled trial with a primary focus on evaluating effectiveness of HealthyTogether and a secondary focus on understanding determinants of implementation. The aims of the trial are:

1. Test whether HealthyTogether results in greater weight loss than usual care at 6 months among Veterans (primary).
2. Examine differences between HealthyTogether and usual care groups in secondary Veteran and partner outcomes, including health behaviors (i.e., diet, physical activity) and relationship quality.
3. Examine Veteran and partner contributions to changes in their own and each other's outcomes using dyadic analyses, informing potential future intervention targets.
4. Assess determinants of implementation, including cost, feasibility, acceptability, and appropriateness, guided by the Consolidated Framework for Implementation Research, to inform future implementation.

Considering the burden of overweight and obesity in VA and the limited reach and effectiveness of MOVE!, HealthyTogether has the potential to address multiple VA priorities: mitigate obesity-related chronic disease and involve family in Veterans' care. Study findings will inform VA National Center Health for Health Promotion and Disease Prevention efforts to expand effective, evidence-based weight management services for Veterans.

ELIGIBILITY:
Inclusion Criteria:

Veteran participants:

* Age 18 or higher.
* Assigned to a VA primary care provider.
* Have a weight measurement (BMI>=30) recorded in the VA medical record within 16 weeks prior to enrollment.
* Have a second, valid weight measurement recorded in the VA medical record within the prior year.
* Have a BMI>=30 at enrollment.
* Able to participate in virtual intervention sessions during regular business hours.

Partner participants:

* Age 18 or higher.
* Able to participate in virtual intervention sessions during regular business hours.
* Speak with Veteran at last weekly.

Exclusion Criteria:

Veterans are excluded if:

* not fluent in English
* have severe hearing loss prohibiting participation
* have a dementia diagnosis
* have recently (within the past 3 months) participated in a clinical or research behavioral weight management program
* have a history of or plans (within 6 months) to have bariatric surgery
* are pregnant, postpartum, nursing, or planning to become pregnant within 6 months
* are receiving cancer (non-skin) treatment
* have drug or alcohol dependence not in remission, a recent suicide attempt, active psychosis, or an active behavior flag in the medical record
* report high-levels of alcohol use (AUDIT-C score >=8)
* are receiving hospice or palliative care
* are living in a nursing home or assisted living facility
* are enrolled in VA home-based primary care
* have end stage renal disease
* have a current or past diagnosis of anorexia or bulimia
* have had an inpatient hospitalization in the past 3 months
* weigh more than 440 pounds (this is the upper limit of the study's scales)

Partners are excluded if:

* not fluent in English
* have severe hearing loss prohibiting participation
* endorse having a health condition that may limit their ability to participate in the intervention
* report high-levels of current alcohol use (AUDIT-C score >=8)
* are receiving hospice or palliative care
* are living in a nursing home or assisted living facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in weight from Baseline to 6-months among Veterans | 6-months
  Weight is measured using a study-provided scale during a scheduled virtual study visit. Veterans will either (1) display the weight on the scale to study staff or (2) take a picture of the weight on the scale with a digital device and show the weight to study staff. For weight measurements at both timepoints, we will instruct participants to weigh themselves in light clothing and no shoes, with the scale on a hard, flat surface. We will record date and time of weight assessments and will make every attempt to collect follow-up weights at a similar time of day as baseline.

SECONDARY OUTCOMES:
Change in weight from Baseline to 6-months among Veterans (including EHR-data) | 6-months
  We will collect supplementary EHR-based weights from for all Veteran participants. We will use the EHR weight closest to 182 days +/- 60 days post-baseline. While the primary outcome is limited to Veterans with study team measured weight, secondary analyses will be conducted among all participants with available weight outcomes (staff verified and/or EHR-based).
Change in weight from Baseline to 6-months among partners | 6-months
  Weight is measured using a study-provided scale during a scheduled virtual study visit. Partners will either (1) display the weight on the scale to study staff or (2) take a picture of the weight on the scale with a digital device and show the weight to study staff. We will record date and time of weight assessments and will make every attempt to collect follow-up weights at a similar time of day as baseline.
Change in weight from Baseline to 12-months among Veterans (using EHR data) | 12-months
  Baseline weight is measured using a study-provided scale during a scheduled virtual study visit. To examine durability of intervention effects while minimizing participant burden, we will also obtain EHR-based weights at 12 months, using weights collected 365 days +/- 90 days post-baseline among only Veterans.
Change in self-reported diet quality from Baseline to 6-months among Veterans | 6-months
  This outcome is measured by self-report using the eight-item Starting the Conversation measure.
Change in self-reported diet quality from Baseline to 6-months among partners | 6-months
  This outcome is measured by self-report using the eight-item Starting the Conversation measure.
Change in physical activity from Baseline to 6-months among Veterans | 6-months
  This outcome is measured by self-report using the 9-item International Physical Activity Questionnaire-Short Form.
Change in physical activity from Baseline to 6-months among partners | 6-months
  This outcome is measured by self-report using the 9-item International Physical Activity Questionnaire-Short Form.
Change in relationship quality from Baseline to 6 months among Veterans | 6-months
  This outcome is assessed by self-report with the seven-item Relationship Assessment Scale, revised for non-romantic relationships.
Change in relationship quality from Baseline to 6 months among partners | 6-months
  This outcome is assessed by self-report with the seven-item Relationship Assessment Scale, revised for non-romantic relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen E. Gray, PhD MS BS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data will be made available outside VA in response to a properly prepared Freedom of Information Act request submitted to the VA Puget Sound FOIA Officer, or submitted and passed down to the facility FOIA Officer from higher VA authority (e.g. VISN 20 or Central Office). Such requests will be evaluated in terms of protecting potential intellectual property value and rights of VA and its employees, collaborators and research sponsors, and any other proprietary or security concerns, including protection of Personal Identifiable Information (PII) and Protected Health Information (PHI), terms of Confidentiality Agreements or other such restrictions and protections.